CLINICAL TRIAL: NCT00963573
Title: Efficacy and Safety of Loratadine-Betamethasone Oral Solution (1 mg/0.05 mg/1 mL) for Initial Treatment of Severe Perennial Allergic Rhinitis in School Age Children
Brief Title: Efficacy & Safety of Loratadine-Betamethasone Oral Solution for Treatment of Severe Perennial Allergic Rhinitis in Children (Study P03428)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P03428
Record Dates: First submitted 2009-08-20; First posted 2009-08-21 (Estimated); Last update posted 2015-04-21 (Estimated); Status verified 2015-04

CONDITIONS: Rhinitis
MeSH Terms: conditions — Rhinitis | interventions — Loratadine; Betamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- loratadine/betamethasone oral solution (Experimental): loratadine/betamethasone oral solution (1 mg/0.05 mg/1 mL), at a dose of 10 mg/0.5 mg
  Interventions: Drug: Loratadine; Drug: Betamethasone

INTERVENTIONS:
Drug: Loratadine — loratadine/betamethasone oral solution (1 mg/0.05 mg/1 mL), at a dose of 10 mg/0.5 mg
  Other Names: SCH 029851
Drug: Betamethasone — loratadine/betamethasone oral solution (1 mg/0.05 mg/1 mL), at a dose of 10 mg/0.5 mg
  Other Names: SCH 029851

SUMMARY:
This study attempts to document the therapeutic value of combining loratadine antihistamine action (no sedative) with anti-inflammatory effects of betamethasone at low doses, which may facilitate treatment adherence by patients whereas providing an effective and rapid perennial allergic rhinitis (PAR) symptoms relief.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of perennial allergic rhinitis.
* Age >= 6 years old and <= 12 years old.
* Patients in good general conditions, without any other relevant clinical condition except for perennial allergic rhinitis.
* Symptoms total score at admission >= 8 (out of 15 possible). Individual symptoms (score 0 to 3 points) were: Sneezing or nasal pruritus, eye reddening or pruritus, nasal congestion, wet nose or with secretion (sniffing), secretion sensation at pharynx (post-nasal dripping).
* Number of symptoms: At least three.

Exclusion Criteria:

* Age < 6 years old or > 12 years old.
* Co-existence of acute sinusitis or some chronic condition different from asthma or atopic dermatitis.
* Presence of systemic fungal infections.
* Conscience or behavioral disturbances.
* Current oral or parenteral steroid treatment.
* Concomitant use of Phenobarbital, rifampicin, diphenylhydantoin or ephedrine.
* Known hypersensitivity to any of the study pharmacological combination components.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2003-09; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
To evaluate efficacy and safety of loratadine/betamethasone oral solution (1 mg/0.05 mg/1 mL), at a dose of 10 mg/0.5 mg, respectively, as an initial treatment for severe perennial allergic rhinitis in school age children | Day 6 (Final visit)

REFERENCES:
- [Result] Mendoza de Morales T, Sanchez F. Clinical efficacy and safety of a combined loratadine-betamethasone oral solution in the treatment of severe pediatric perennial allergic rhinitis. World Allergy Organ J. 2009 Apr;2(4):49-53. doi: 10.1097/WOX.0b013e31819f2105. PMID 23282980